CLINICAL TRIAL: NCT05137015
Title: Preventing Injuries in Young Football Players: a Cluster Randomised Controlled Trial
Brief Title: Preventing Injuries in Young Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Injury Prevention Study 21/22
Record Dates: First submitted 2021-11-18; First posted 2021-11-30 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Injury Prevention

STUDY DESIGN:
Intervention Model Description: Cluster randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: Two teams will work on injury data collection. Teams are not informed for which group (intervention or control) they are recording the datas.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will use the new injury prevention program at least twice per week in their training sessions.
  Interventions: Other: Injury prevention program
- Control (No Intervention): The control group will continue their usual training routine.

INTERVENTIONS:
Other: Injury prevention program — The execution of the program takes 10-15 minutes. The program will be performed in the training sessions, after the usual warm-up.
  The program is based on scientific evidence that has previously shown good efficacy on injury prevention in football. The exercise categories address 7 aspects:
  1. Balance
  2. Core stability
  3. Hamstring eccentrics
  4. Glute activation
  5. Plyometrics
  6. Running
  7. Games The games are included with the aim to increase the attractiveness of the program.
  Each category contains 2 exercises and the coach is free to decide which one to choose in every training session. All exercises are organized in five or six levels with increasing difficulty (physically and cognitively).
  Arms: Intervention

SUMMARY:
Football is the most popular sport in the world, with 260 million male and female active participants, including ~113,000 FIFA registered professional players. Playing football is fun and can provide many health benefits, however, it also presents a high injury risk. Studies on elite and non-elite footballers have reported similar injury rates in both genders. The most common football-related injuries are the knee and ankle ligament and thigh muscle strains, Over the past two decades, significant advancement has been made in the field of injury prevention in football. There are used trials to prevent specific injuries, as ankle sprain, ACL injuries, hamstring strains, etc. On the other hand, there are created programs designed to prevent a wider spectrum of injuries like FIFA11+.

Therefore, the aim of this study is to investigate the effect of a new injury prevention program on the overall injury incidence in young football players.

ELIGIBILITY:
Inclusion Criteria:

officially registered football club in the football federation of Kosovo players must be between 13-19 years old regular training must take place at least three times per week

Exclusion Criteria:

teams already using an injury prevention program injured players

Ages: 13 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1027 (Actual)
Dates: Start 2021-09-04 (Actual); Primary Completion 2022-05-29 (Actual); Study Completion 2023-01-21 (Actual)

PRIMARY OUTCOMES:
Overall injury rate | up to 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Gjakova, Gjakova, Kosovo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Obertinca R, Meha R, Hoxha I, Shabani B, Meyer T, Aus der Funten K. Impact of the 'FUNBALL' Programme on Severe Injuries Among Young Male Football Players: A Secondary Analysis from a Cluster-Randomised Controlled Trial. Sports Med Open. 2025 Nov 27;11(1):151. doi: 10.1186/s40798-025-00945-3. PMID 41310111
- [Derived] Obertinca R, Meha R, Hoxha I, Shabani B, Meyer T, Aus der Funten K. Efficacy of a new injury prevention programme (FUNBALL) in young male football (soccer) players: a cluster-randomised controlled trial. Br J Sports Med. 2024 May 2;58(10):548-555. doi: 10.1136/bjsports-2023-107388. PMID 38499320